CLINICAL TRIAL: NCT02672930
Title: How Much Reliable iv Calcium for the Treatment of Hyperkalemia?
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Adnan Yamanoğlu, Emergency Medicine Specialist, Haseki Training and Research Hospital
Other Study IDs: 230
Record Dates: First submitted 2016-01-17; First posted 2016-02-03 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2020-09

CONDITIONS: Acute Renal Failure; Chronic Renal Failure
Keywords: calcium gluconate; hyperpotassemia treatment
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Electrocardiogram (ECG) — ECG and vital parameters were obtained before and after recommended standard calcium gluconate therapy for hyperkalemia

SUMMARY:
Hyperkalemia is a common problem in the emergency services and one of the life threatening metabolic emergencies. Calcium, insulin, beta adrenoceptor agonists, bicarbonate, diuretics, sodium polystyrene sulfonate and lastly dialysis are advised in treatment. Especially, avoiding evolution of serious arrythmias and iv calcium using in the treatment of occured electrocardiogram (ECG) abnormalities, there is not sufficient level of survey in the literature. So the aim of this study was to evaluate administration of iv calcium efficiency on vital signs and ECG.

DETAILED DESCRIPTION:
Hyperkalemia is a common problem in the emergency services and one of the life threatening metabolic emergencies. Serious hyperkalemia is mostly seen in patients who have known chronic renal failure or end stage renal disease, and also new diagnosis of acute renal failure can be appear with serious hyperkalemia. Paresthesia and weakness which is proceeded to flask paralysis can be observable, sharp ''T'' waves (the repolarization and relaxation of the ventricles), diminution of ''P'' waves (atrial depolarisation and contraction), long ''PR'' intervals (time frame from the beginning of atrial depolarization to the beginning of ventricular depolarization), or elongated ''QRS'' complexes (depolarisation and contraction of the ventricles), ''ST'' segment (end of the QRS complex to the beginning of the T wave) elevation, and serious ventricular arrythmias can be seen in electrocardiography. Calcium, insulin, beta adrenoceptor agonists, bicarbonate, diuretics, sodium polystyrene sulfonate and lastly dialysis are advised in treatment. Especially, avoiding evolution of serious arrythmias and İv calcium using in the treatment of occured ''ECG'' abnormalities, there is not sufficient level of survey in the literature. The group of Cochrane stated in systematic assessment report, which is published in 2005 about IV calcium administration, available dates are based on anecdotal and animal experiments. And in the researches that we have done, we did not find clinical human studies showing the benefits of calcium administration beyond the delivery of case reports . The aim of this study was to evaluate administration of İv calcium efficiency on vital signs and ECG.

ELIGIBILITY:
Inclusion Criteria:

* All patients who had ECG changes due to hyperpotassemia (K>5.5 mmol/l)

Exclusion Criteria:

* Arrest patients
* Patients needed antiarrhythmic interventions
* Patients need inotropic that may cause ECG changes
* Patients need atropine during emergency treatment prior to Ca-gluconate
* Patients needed cardioversion or defibrillation
* Hyperpotassemia with myocardial infarction
* In the presence of other situations which changes ECG for example pericarditis
* Unstabile patients for ideal ECG
* Digoxin usage
* Trauma
* blood calcium level of > 10.5 mg/dl

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Blood potassium levels above 5.5 and all patients with ECG changes due hyperpotassemia were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
ECG changes after the calcium infusion | 10 minutes

SECONDARY OUTCOMES:
Pulse changes after the calcium infusion | 10 minutes
Blood pressure changes after the calcium infusion | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Yamanoğlu, MD, Principal Investigator — Emergency Department
Locations (1):
- Haseki Training and Reseurch Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No